CLINICAL TRIAL: NCT02790619
Title: A Pilot Study Investigating Transcranial Direct Current Stimulation (tDCS) to Enhance Mindfulness Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00042149
Record Dates: First submitted 2015-07-13; First posted 2016-06-06 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meditation and Active Stimulation 1 (Active Comparator): Electrodes will then be placed on the participant and participant will then listen to a meditative recording instructing to focus on participant's breath that will last approximately 5 minutes.Participant will then receive 20 minutes of tDCS with Anode over F8 and cathode over left supraorbital area with 1 milliamp(mA) stimulation with intervention administration delivered by tDCS via Chattanooga Ionto Iontophoresis System-Phoresor.
  Interventions: Device: tDCS via Chattanooga Ionto Iontophoresis System-Phoresor
- Meditation and Active Stimulation 2 (Active Comparator): Electrodes will then be placed on the participant and participant will then listen to a meditative recording instructing to focus on participant's breath that will last approximately 5 minutes.Participant will then receive 20 minutes of tDCS with Anode over F8 and cathode over left supraorbital area with 2 mA stimulation with intervention administration delivered by tDCS via Chattanooga Ionto Iontophoresis System-Phoresor.
  Interventions: Device: tDCS via Chattanooga Ionto Iontophoresis System-Phoresor
- Meditation and Sham Stimulation (Sham Comparator): Electrodes will then be placed on the participant and participant will then listen to a meditative recording instructing to focus on participant's breath that will last approximately 5 minutes.The participants in the sham study will receive Sham tDCS (no stimulation) with Anode over F8 and cathode over left supraorbital area with intervention administration delivered by Sham tDCS Chattanooga Ionto Iontophoresis System-Phoresor
  Interventions: Device: Sham tDCS Chattanooga Ionto Iontophoresis System-Phoresor

INTERVENTIONS:
Device: tDCS via Chattanooga Ionto Iontophoresis System-Phoresor — Small electrical current delivered non-invasively to the scalp. 1mA electrical current to Meditation and Active Stimulation 1 condition. 2mA to Meditation and Active 2 Stimulation condition.
  Arms: Meditation and Active Stimulation 1; Meditation and Active Stimulation 2
Device: Sham tDCS Chattanooga Ionto Iontophoresis System-Phoresor — Blinds participants to meditation condition by applying 30 seconds of real stimulation and then turning the device off.
  Arms: Meditation and Sham Stimulation

SUMMARY:
The purpose of this study is to determine if a new technology applied while listening to a mindfulness meditation tape can affect one's ability to achieve a state of "mindfulness." The new technology is called transcranial direct current stimulation, or tDCS.

DETAILED DESCRIPTION:
Many people initially attempt meditation but cannot get their mind to be still. Or they do not get quick results and find it frustrating. Thus, the number of people benefiting from meditation would increase if there were a method of making it easier to perform. Moreover, establishing the actual brain mechanisms involved in the benefits of meditation would potentially open up synergistic treatments and approaches.

The investigators will investigate the use of a new, non-invasive brain stimulation method called transcranial direct current stimulation (tDCS) to augment a state of mindfulness. tDCS is a safe, inexpensive, non-invasive brain stimulation modality that has the capability of focally increasing or decreasing cortical activity. Anodal stimulation produces positive DC stimulation and is associated with increased cortical activity, whereas Cathodal stimulation produces a negative DC stimulation and is associated with decreased cortical activity. Cortical activity changes occur both during and after stimulation in a dose response fashion (higher current density and longer duration of stimulation produces larger and longer lasting effects).

The investigators will be investigating the use of tDCS to augment mindfulness meditation in a double-blind, crossover, randomized, sham-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control volunteers.
* meditation naive

Exclusion Criteria:

* Pregnancy,
* History of Mental illness or neurological disorders,
* prior meditative experiences

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Mood Visual Analog Scale (Mood VAS) at Post Stimulation of Experimental Visit One | Baseline (Visit 1/Week 1) Post Stimulation (Visit 1/Week 1). Through Visit 1 completion, an average of 25 minutes
  During Experimental Visit 1 the participant will complete the Mood Visual Analog Scale before listening to a meditative tape recording and receiving either active tDCS or sham tDCS for 20 minutes. The participant will then fill out the Mood Visual Analog Scale post stimulation.
Change from Baseline Mood Visual Analog Scale (Mood VAS) at Post Stimulation of Experimental Visit Two | Baseline (Visit 2/Week 2) Post Stimulation (Visit 2/Week 2). Through Visit 2 completion, an average of 25 minutes
  During Experimental Visit 2 the participant will complete the Mood Visual Analog Scale before listening to a meditative tape recording and receiving either active tDCS or sham tDCS for 20 minutes. The participant will then fill out the Mood Visual Analog Scale post stimulation.
Change from Baseline Mood Visual Analog Scale (Mood VAS) at Post Stimulation of Experimental Visit Three | Baseline (Visit 3/Week 3) Post Stimulation (Visit 3/Week 3). Through Visit 3 completion, an average of 25 minutes
  During Experimental Visit 3 the participant will complete the Mood Visual Analog Scale before listening to a meditative tape recording and receiving either active tDCS or sham tDCS for 20 minutes. The participant will then fill out the Mood Visual Analog Scale post stimulation.